CLINICAL TRIAL: NCT06040567
Title: Polyneuropathy, Impairments and Physical Activity - The PolyImPAct Study
Acronym: PolyImPAct
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Britt Stævnsbo Pedersen, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: H-23032160
Record Dates: First submitted 2023-09-01; First posted 2023-09-15 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy (CIDP); Vasculitic Neuropathy; POEMS Syndrome; Multifocal Motor Neuropathy; Charcot-Marie-Tooth; hATTR Amyloidosis; Diabetic Polyneuropathy; Idiopathic Neuropathy; Polyneuropathies
Keywords: Polyneuropathy; Clinical outcome measures; Patient reported outcome measures (PROMs); Physical activity; Accelerometer; Validity; Reliability; Responsiveness
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; POEMS Syndrome; Charcot-Marie-Tooth Disease; Diabetic Neuropathies; Polyneuropathies; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with polyneuropathy: Adults (> 18 years) diagnosed with polyneuropathy
  Interventions: Other: Validity and reliability of outcome measures in polyneuropathy
- Healthy controls: Healthy adults (>18 years)
  Interventions: Other: Healthy controls

INTERVENTIONS:
Other: Validity and reliability of outcome measures in polyneuropathy — Patients will be tested, answer patient reported outcome measures, and wear accelerometer at baseline after 2-4 weeks and after 1-2 years.
  Groups: Patients with polyneuropathy
Other: Healthy controls — Healthy controls will be tested, answer patient reported outcome measures, and wear accelerometer at baseline visit. There is no follow-up in the healthy control group.
  Groups: Healthy controls

SUMMARY:
The project aims to investigate the validity, and reliability of outcome measures of muscle strength, functioning (gait, balance, and fine motor skills), physical activity, and patient-reported outcome measures of functioning (gait, balance, and fine motor skills), and daily living among patients with polyneuropathy. Further, the project aims to compare physical activity and patient-reported outcome measures of functioning (gait, balance, and fine motor skills), and daily living among patients with polyneuropathy with physical activity and patient-reported outcome measures of functioning (gait, balance, and fine motor skills) and daily living in healthy adults.

DETAILED DESCRIPTION:
In four phases the investigators will evaluate physical activity and the validity, reliability, and responsiveness of the outcome measures in patients with polyneuropathy. During the four phases clinical outcome measures, patient-reported outcomes measures, and accelerometer data on physical activity will be evaluated. The investigators plan to include 400 adult patients with polyneuropathy (acquired, hereditary, and idiopathic) from our clinic and 120 adult healthy controls. The 400 patients with polyneuropathy include the following subtypes of polyneuropathy: Chronic Inflammatory Demyelinating Polyneuropathy (CIDP), vasculitis polyneuropathy, Polyneuropathy-Organomegaly-Endocrinopathy-Monoclonal protein-Skin changes (POEMS syndrome), Multifocal Motor Neuropathy (MMN), Charcot Marie Tooth (CMT), hATTR amyloidosis, Diabetic Polyneuropathy (DPN), and idiopathic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria patients:

> 18 years Diagnosed with polyneuropathy (verified by nerve conduction)

Inclusion Criteria healthy controls:

> 18 years Healthy

Exclusion Criteria:

Exclusion Criteria patients:

Not verified polyneuropathy

Exclusion Criteria healthy controls:

Diabetes, brain-, nerve-, muscle-, kidney-, or liver disease. Diagnosed with polyneuropathy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from a the neuromuscular clinic at Rigshopitalet, Copenjagen, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2023-09-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
10-meter Walk Test | At baseline (study entry), after 2-4 weeks, and after 1-2 years
  The patient is asked to 10 meter as fast as possible
Six Spot Step Test | At baseline (study entry), after 2-4 weeks, and after 1-2 years
  The patient is instructed to walk 5 meters as fast as possible, while kicking five cylinder blocks out of five circles marked on the floor.
6-minute Walk Test | At baseline (study entry), after 2-4 weeks, and after 1-2 years
  The patient will be asked to walk back and forth along a 25 meter walkway for six minutes. They will be instructed to walk as far as possible for six minutes.
30 seconds Chair Stand Test | At baseline (study entry), after 2-4 weeks, and after 1-2 years
  The patients will be asked to stand up and sit down as many times as possible in 30 secs with their arms across their chest
Dynamic Gait Index | At baseline, after 2-4 weeks, and after 1-2 years
  The patient will be asked to walk while performing different tasks (walking: normally, while changing speed, while turning head (vertical and horizontal), while turning around, while stepping over obstacles, and walking stairs).
Nine Hole Peg Test | At baseline (study entry), after 2-4 weeks, and after 1-2 years
  Fine motor skills
Jamar Hand-grip dynamometer (hand-grip-strength) | At baseline (study entry), after 2-4 weeks, and after 1-2 years
  Best of three values
Isometric strength measured with hand-held dynamometer | At baseline (study entry), after 2-4 weeks, and after 1-2 years
  Will be tested bilateral at ankle, knee, wrist and elbow
Isokinetic muscle strength measured with Biodex System 3 or 4 PRO, Biodex Medical Systems | At baseline (study entry), after 2-4 weeks, and after 1-2 years
  Will be tested bilateral at ankle and knee
SENS motion activity sensor (accelerometer) | At baseline (study entry), and after 1-2 years
  The SENS motion activity sensor is a wearable accelerometer. It measures physical activity by collecting raw data of accelerations. Data on active time, sedentary time, time spent walking and number of steps taken will be collected.
  The sensor will be attached and worn 24/7 (the sensor will be worn the week following baseline tests, and the week after tests at visit three (1-2 years after baseline).
Inflammatory Neuropathy Cause and Treatment (INCAT) | At baseline (study entry), after 2-4 weeks, and after 1-2 years
  Interview based disability scale INCAT evaluates disability of the upper and lower limb. The total INCAT score ranges from 0-10 (low scores indicating no disability and higher scores indicating higher level of disability).

SECONDARY OUTCOMES:
Rasch-build Overall Disability Scale for Immune-mediated peripheral neuropathies (I-RODS) | At baseline (study entry), after 2-4 weeks, and after 1-2 years
  I-RODS is a 24-item patient reported outcome measure that measures disability. The raw score ranges from 0-48, with 0 indicating severe disability and higher scores indicating lower levels of disability.
Falls Efficacy Scale-International (FES-I) | At baseline (study entry), after 2-4 weeks, and after 1-2 years
  Assesses limitations related to fear of falling. FES-I is a 16-item patient reported outcome measure that measures fear of falling. The score ranges from 16-64, with higher scores indicating greater fear of falling.
Composite Autonomic Symptom Score (COMPAS-31) | At baseline (study entry), after 2-4 weeks, and after 1-2 years
  Assesses autonomic dysfunction Compass-31 is a patient reported outcome measure that measures autonomic dysfunction. Scores ranges from 0-100, with higher scores indicating more severe symptoms of autonomic dysfunction.
Self-reported Leeds Assessment of Neuropathic Symptoms and Signs (S-LANNS) | At baseline (study entry), after 2-4 weeks, and after 1-2 years
  Assesses neuropathic pain S-LANSS is a patient reported outcome measure for identifying neuropathic pain.
Fatigue Severity Scale (FSS) | At baseline (study entry), after 2-4 weeks, and after 1-2 years
  Assesses fatigue FSS is a 9-item patient reported outcome measure that measures fatigue, and the impact of fatigue on physical activity and daily living. The score ranges from 9-63, with a higher score indicating higher levels of fatigue.
PittsburghSleep Quality Index | At baseline (study entry), after 2-4 weeks, and after 1-2 years
  PittsburghSleep Quality Index is a patient reported outcome measure that assesses sleep quality. The score ranges from 0-21, with higher scores indicating more affected sleep quality
Major Depression Inventory (MDI) | At baseline (study entry), after 2-4 weeks, and after 1-2 years
  MDI is a patient reported outcome measure that measures depressive symptoms. The score ranges from 0-50, with higher scores indicating deeper depression.
International Physical Activity Questionaire (IPAQ) | At baseline (study entry), after 2-4 weeks, and after 1-2 years
  International Physical Activity Questionaire (IPAQ) is a patient reported outcome measure that measures physical activity.
Physical Activity Scale (PAS2) | At baseline (study entry), after 2-4 weeks, and after 1-2 years
  PAS2 is a 7-item patient reported outcome measure that measures physical activity and sedentary behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Britt S Pedersen, Study Chair — Rigshospitalet, University of Copenhagen
Locations (1):
- Copenhagen Neuromuscular Center, Rigshospitalet, Copenhagen, Denmark